CLINICAL TRIAL: NCT01030445
Title: A Pilot Study: Cardiac Function as Measured by Non-invasive Electrical Velocimetry Cardiac Monitor in Hospitalized Children From Acute Illness (Disease) to Recovery (Health).
Brief Title: Cardiac Function as Measured by Non-invasive Electrical Velocimetry Cardiac Monitor in Hospitalized Children
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Jackson Wong, Associate Professor of Pediatrics, Boston Children's Hospital
Other Study IDs: 09-11-0597
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2011-06

CONDITIONS: Cardiac Output; Blood Pressure
Keywords: non-invasive cardiac output monitor; electrical velocimetry; Aesculon; Icon; pediatrics; normal reference

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Elevated Mean Arterial Blood Pressure: Mean arterial pressure greater than 1 standard deviation above the mean based on age
- Decrease Mean Arterial Blood Pressure: Mean arterial pressure greater than 1 standard deviation below the mean based on age
- Normal Mean Arterial Blood Pressure: Mean arterial pressure within the standard deviation of the mean based on age

SUMMARY:
To assess whether a non-invasive cardiac output monitor can follow heart function in children during treatments in the hospital. To establish a normal reference for children who are well and awake.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the ability of a new FDA-approved non-invasive Electrical Velocimetry (EV) cardiac monitor called AESCULON (Cardiotronic Inc, La Jolla CA) to detect and trend hemodynamic changes in hospitalized ambulatory pediatric patients during recovery from acute illness. We postulate that if the cardiac monitor can trend hemodynamic changes in hypertensive patients whose mean arterial pressure (MAP) decreases to normal levels, or hypotensive patients whose MAP increases to normal levels over several days, it may improve our understanding of different disease processes and allow us to improve care. We also seek to establish normative data for different measures provided by the AESCULON monitor - specifically cardiac output (CO) and systemic vascular resistance (SVR), which are the prime determinants of MAP.

ELIGIBILITY:
Inclusion Criteria:

* Medical patients without complex medical history with expected hospital stay for less than 10 days
* Uncomplicated Medical Patients as define as (1) Previously healthy children or (2) Children with diagnosis of a single chronic medical disorder that is not associated with cardiac dysfunction

Exclusion Criteria:

* Congenital heart disease with and without repair (includes PFO, ASD and PDA, cardiac valve disease or pulmonary hypertension
* Chronic lung disease (except asthma)
* Abnormal Hemoglobin (SSD)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized children
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2009-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To document trends in cardiac output (CO) and systemic vascular resistance (SVR) in subjects undergoing systematic changes in mean arterial pressure (MAP) and to assess intra-individual variability for those with normal blood pressure | During hospitalization until discharge

SECONDARY OUTCOMES:
To establish age relevant hemodynamic norms as measured by the electrical velocimetry (EV) cardiac monitor for trend parameters | Measurements obtain on day of discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States